CLINICAL TRIAL: NCT00353015
Title: A Phase II Study of Irinotecan and Cisplatin for Metastatic or Unresectable High Grade Neuroendocrine Carcinoma of the Gastrointestinal Tract
Brief Title: Irinotecan and Cisplatin for High Grade Neuroendocrine Carcinoma of the Gastrointestinal Tract
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Pharmacia (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ID02-523
Record Dates: First submitted 2006-07-13; First posted 2006-07-17 (Estimated); Last update posted 2012-08-02 (Estimated); Status verified 2012-08

CONDITIONS: Gastrointestinal Cancer; Carcinoma, Neuroendocrine
Keywords: Gastrointestinal cancer; high grade gastrointestinal neuroendocrine carcinoma; High grade neuroendocrine carcinoma of unknown primary site; Cisplatin; Platinol-AQ; Platinol; CDDP; CPT-11; Irinotecan
MeSH Terms: conditions — Gastrointestinal Neoplasms; Carcinoma, Neuroendocrine | interventions — Cisplatin; Irinotecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Irinotecan plus Cisplatin (Experimental): Irinotecan 65 mg/m2 and Cisplatin 25 mg/m2 intravenous (IV) days 1, 8 of a 21-day cycle
  Interventions: Drug: Cisplatin; Drug: Irinotecan

INTERVENTIONS:
Drug: Cisplatin — Cisplatin 25 mg/m2 IV days 1, 8 of a 21-day cycle
  Other Names: Platinol-AQ; Platinol; CDDP
Drug: Irinotecan — Irinotecan 65 mg/m2 IV days 1, 8 of a 21-day cycle
  Other Names: CPT-11

SUMMARY:
Primary Objective:

1. Assess the clinical activity defined by response rate of irinotecan and cisplatin in untreated patients with metastatic or unresectable high grade neuroendocrine carcinoma of the gastrointestinal tract.

Secondary Objective:

1. To assess the safety profile of irinotecan and cisplatin in untreated patients with metastatic or unresectable high grade neuroendocrine carcinoma of the gastrointestinal tract.

DETAILED DESCRIPTION:
Both irinotecan and carboplatin are drugs commonly used to treat cancer.

Before treatment starts, patients will have blood tests (around 4 teaspoons) and urine tests. Patients will have a chest X-ray, an electrocardiogram (ECG-a test to measure the electrical activity of the heart), and a computed tomography (CT) scan. Women who are able to have children must have a negative blood pregnancy test.

During the study, patients will receive irinotecan and cisplatin by vein over 4 hours, once a week for 2 weeks. This will be followed by 7 days in which no treatment will be given. This 3 week period is called a cycle. Cycles will be repeated unless the tumor continues to grow.

During treatment, patients will have follow-up visits every 3 weeks to check for any side effects and the status of the disease. The follow-up visits may be with either your local doctor or with the study doctor. However, visits with the study doctor should be scheduled at least every 9 weeks. If the disease gets worse or you experience any intolerable side effects, you will be taken off the study.

This is an investigational study. Both irinotecan and cisplatin are FDA approved and commercially available. Around 36 patients will participate in the study. All patients will be enrolled at M.D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Histologic diagnosis of high grade (poorly differentiated, small cell) gastrointestinal neuroendocrine carcinoma.
2. High grade neuroendocrine carcinoma of unknown primary site (if a pulmonary primary has been excluded).
3. Metastatic or unresectable disease.
4. Measurable disease.
5. Informed consent.
6. Zubrod performance status of 0 or 1.
7. Adequate bone marrow function (defined as absolute neutrophil count [ANC] >= 1500, platelet count [PLT] >= 100,000 and a hemoglobin [Hgb] >= 10).
8. Adequate hepatic function with a bilirubin of <= 2.0 mg/dl, and aspartate aminotransferase (AST or SGOT) and alanine aminotransferase (ALT or SGPT) <= 2.5 times the upper limits of normal, unless caused by liver metastasis. If caused by metastasis, then should be SGPT and SGOT <= 5 times the upper limits of normal.
9. Adequate renal function defined as serum creatinine <= 1.5 mg/dl.
10. Fertile patients and their partners must practice appropriate contraceptive methods while on study.
11. Recovered from recent surgery. One week must have elapsed from the time of a minor surgery and 3 weeks from major surgery.

Exclusion Criteria:

1. Patients with prior systemic chemotherapy are ineligible.
2. Other concurrent chemotherapy, immunotherapy, or radiotherapy.
3. Patients with brain metastases are not eligible. Patients with a history of seizures are ineligible. Patients receiving phenytoin, phenobarbital, or other antiepileptic prophylaxis are ineligible.
4. Patients with New York Heart Association (NYHA) Class III or IV heart disease are not eligible as well as those patients with history of angina, myocardial infarction, or congestive heart failure within six months.
5. Pregnant or lactating women. All women of child bearing potential must have a negative pregnancy test prior to entry into the study. All patients of child bearing potential must be advised of the importance of avoiding pregnancy and using appropriate methods of contraception while participating in this investigational trial.
6. Patients with serious intercurrent infections, or nonmalignant medical illnesses that are uncontrolled or whose control may be jeopardized by the complications of this therapy, are ineligible.
7. Patients with psychiatric disorders rendering them incapable of complying with the requirements of the protocol are ineligible.
8. Patients with serum calcium > 12 mg/dl or symptomatic hypercalcemia under treatment are ineligible.
9. Patients with osseous metastasis as only site of disease.
10. Patients with any concurrent active malignancy other than non-melanoma skin cancers or carcinoma-in-situ of the cervix. Patients with previous malignancies but without evidence of disease for > 5 years will be allowed to enter the trial.
11. Patients with known Gilbert's syndrome are ineligible.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2003-03; Primary Completion 2007-12 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
Participant Response Rate of Irinotecan and Cisplatin | Every 3 weeks
  Clinical activity defined by number of participants with Complete Response (CR) and Partial Response (PR) divided by total number of particpants using Response Evaluation Criteria in Solid Tumors (RECIST) where changes in tumor measurements confirmed by repeat assessments no less than 4 weeks after criteria for CR and PR responses first met.

CONTACTS AND LOCATIONS:
Overall Officials: James C. Yao, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- U.T. M.D. Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: The University of Texas M.D.Anderson Cancer Center — http://www.mdanderson.org